CLINICAL TRIAL: NCT04620356
Title: Effect of Use of DryNites Absorbent Pants on the Rate of Spontaneous Resolution of Paediatric Nocturnal Enuresis (NE)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kimberly-Clark Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KCC-DN-001
Record Dates: First submitted 2020-09-23; First posted 2020-11-09 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Nocturnal Enuresis
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DryNites arm (Experimental): Participants in this arm use DryNites every night for 4 weeks ("run-in" period), an additional 4 weeks (intervention "core trial" period), and an optional additional 4 weeks ("extension" period). All participants in this arm also receive absorbent bad mats to use every night.
  Interventions: Device: DryNites Pyjama Pants
- No Pants arm (No Intervention): Participants in this arm use DryNites every night for 4 weeks only during the initial "run-in" period. Thereafter, participants in this arm do not use DryNites during the 4 week intervention "core trial" period or the optional additional 4 weeks "extension" period. All participants in this arm also receive absorbent bad mats to use every night.

INTERVENTIONS:
Device: DryNites Pyjama Pants — DryNites Pyjama Pants are disposable, absorbent youth pants designed to help children manage bed wetting by absorbing involuntary urine loss and protecting the child's garments and bedding. DryNites Pyjama Pants are underwear-like alternatives that can be discreetly worn beneath pyjamas or nightwear during the bedwetting phase.
  Arms: DryNites arm

SUMMARY:
Children vary in the age at which they achieve night-time dryness; in almost all cases children will stop bed-wetting without any need for treatment. Use of absorbent pants for the management of nocturnal enuresis is controversial regarding the impact on the speed at which children become dry throughout the night. The aim of this study is to determine the effect of using DryNites absorbent pants in children with monosymptomatic nocturnal enuresis on the speed they become dry throughout the night compared with removing absorbent pants.

DETAILED DESCRIPTION:
Children with severe monosymptomatic NE between 4 and 8 years of age were recruited from study centers in Denmark, Belgium, and the UK. All participants had used absorbents pandt of any manufacturer for at least the previous 6 months. Participants fulfilling the inclusion criteria entered a 4-week run-in period during which they slept wearing the intervention absorbent pant. To be eligible for randomization, participants needed to have 7/7 wet nights in the last week of the run-in period. Eligible participants were then randomly assigned (2:1) to either discontinuation or continuation of absorbent pants for the 4-week core intervention period. The children sleeping without absorbent pants were permitted to sleep with an absorbent bed mat instead. No behavioral changes such as fluid restriction or lifting the child to the toilet when the parents went to bed were allowed in either group. After completing the core intervention period, participants were invited to take part in a 4-week extension period, during which they would remain on their randomly assigned treatment. Number of wet nights were assesed during the study using an electronic diary. Quality- of- life (QoL) and sleep parameters were assessed using the following validated questionnaires: Paediatric Incontinence Questionnaire (PinQ), World Health Organization Quality of Life Brief Version Paediatric Daytime Sleepiness Scale (PDSS), and Checklist Individual Strength. Questionnaires were completed jointly by children and parents.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 4-8 years at the time of enrollment
* Have a clinical diagnosis of monosymptomatic primary NE
* Have been dry in the day for >/= 6 months prior to enrollment
* Have on average no more than 1 dry night per month during the past 6 months at enrollment
* Have an informed consent signed by the their parent(s)/carer(s)

Exclusion Criteria:

* Children in foster/court care
* Have implemented any previous intervention to address NE (use of prescribed alarm schedule, desmopressin, imipramine, anticholinergics) or withdrawal of pants/nappies for > 7 days in the previous 6 months
* Have secondary NE
* Have wetting in the day
* Have faecal soiling
* Have known urinary tract disease
* Have diabetes
* Receive any regular intake of medication
* Have a known developmental/neurological disorder
* Have links to Kimberly-Clark of any kind (including family relations employed by Kimberly-Clark, holding stocks or share in Kimberly-Clark)

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2023-01-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren Riting, Principal Investigator — Department of Pediatrics, Aarhus University Hospital, Aarhus, Denmark
Locations (2):
- United Kingdom (2):
  - Mounts Bay Medical, Connor, Haley
  - Siddarth Marnekar, Hull

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breinbjerg A, Kamperis K, Thorsteinsson K, Jorgensen CS, Dossche L, Rayner J, Zhang J, Rodrigues DG, Borch L, Hagstrom S, Tekgul S, Walle JV, Rittig S. Discontinuing absorbent pants in children with bedwetting: a randomized controlled trial. Eur J Pediatr. 2024 May;183(5):2443-2453. doi: 10.1007/s00431-024-05502-w. Epub 2024 Mar 12. PMID 38472381

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited both from the community and from primary and tertiary care centers.
Pre-assignment Details: Assessed for eligibility (n = 116). Excluded pré randomization(n = 11)
  * Not meeting inclusion criteria (n = 1)
  * Not meeting randomisation criteria (n = 9)
  * Severe non-compliance (n = 1)
Period: Overall Study
Arm/Group | DryNites Arm | No Pants Arm
Started | 35 | 70
Completed | 31 | 49
Not Completed | 4 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DryNites Arm | No Pants Arm | Total
Number analyzed (Participants) | 35 | 70 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (1.22) | 5.6 (1.09) | 5.6 (1.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 29 | 43
  Male | 21 | 41 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 69 | 104
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 35 | 70 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Wet Nights
Description: Average number of wet nights
Time Frame: Last week of the 4-week intervention period
Measure: Mean (Standard Deviation); unit: wet nights per week
Arm/Group | DryNites Arm | No Pants Arm
Number analyzed (Participants) | 34 | 66
wet nights per week | 2.4 (2.21) | 4.6 (1.99)

2. Secondary Outcome: Impact of Urinary Incontinence on Emotional Wellbeing of Child as Assessed by Paediatric Incontinence Questionnaire (PinQ)
Description: The PinQ will be used to assess the child's QoL. The PinQ is a validated cross-cultural continence-specific paediatric QoL questionnaire to assess children with bladder dysfunction, developed by Bower el al (Bower et al. 2006). It is available as self-rated and proxy versions.
  This will be completed by the child themselves in the older participant group and will be completed by the parent/carer on behalf of the child in the younger participant group.
  The PinQ measures the emotional impact that urinary incontinence has on a child. It consists of 20 urinary incontinence QoL related questions divided in 2 dimensions: intrinsic (14 items) and extrinsic (6 items), which are graded on a scale of 0 to 4 (0=No, 1=Hardly ever,2=Sometimes, 3=Often, 4=All the time) with a score range of 0 to 80.
  The total score indicates the impact urinary incontinence has on the child's QoL with the higher scores indicating a more significant effect.
Time Frame: Assessment will be done at each study clinic visit (Day 56 +/- 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DryNites Arm | No Pants Arm
Number analyzed (Participants) | 29 | 58
score on a scale | 12.9 (8.17) | 15.2 (10.83)

3. Secondary Outcome: Impact of Child Nighttime Enuresis on Parent/Carer Quality of Life as Assessed by the WHOQoL-BREF Questionnaire
Description: The WHOQoL-BREF questionnaire (WHO 1996) will be completed directly by the parent/carer. . The WHOQoL-BREF questionnaire is derived from a larger instrument, the WHOQoL-100. It includes 26 items, grouped in 4 domains: Physical Heath, Psychological, Social Relationships, and Environment, and 2 separate items asking the crespondent about overall perception of QoL (item 1) and an individual's overall perception of their health (item 2). The scores of items 3, 4 and 5, which are negatively phrased, need to be reversed. The mean score of items within each domain is used to calculate the domain scores, which are converted into a 0-100 scale. Higher scores denote higher QoL. Where more than 20% of data is missing from an assessment, the assessment should be discarded. Where an item is missing, the mean of other items in the domain is substituted. Where more than 2 items are missing from the domain, the domain score should not be calculated
Time Frame: Assessment will be done at each study clinic visit (Day 56 +/- 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DryNites Arm | No Pants Arm
Number analyzed (Participants) | 29 | 62
score on a scale | 21.3 (3.13) | 21.5 (3.86)

4. Secondary Outcome: Child Daytime Sleepiness as Assessed by PDSS Questionnaire
Description: The Paeditric Daytime Sleepiness Scale (PDSS) questionnaire measures daytime sleepiness in children. It is comprised of 8 items assessing daytime sleepiness and rated on a 5-point scale with 0 = Never and 4 = Always/Very Often. The scale ranges from 0 to 32. The questionnaire will be completed by the child themselves (with attendance of an adult) in the older participant group and by the parent/carer on behalf of the child in the younger participant group. Higher scores indicate greater daytime sleepiness. Higher scores indicate greater daytime sleepiness, and were associated with reduced total sleep time, poorer school achievement, poorer anger control, and frequent illness.
Time Frame: Assessment will be done at each study clinic visit (Day 56 +/- 7)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DryNites Arm | No Pants Arm
Number analyzed (Participants) | 32 | 61
score on a scale | 7.7 (3.63) | 8.5 (4.13)

5. Secondary Outcome: Parent/Carer Fatigue as Assessed by Checklist Individual Strength (CIS Questionnaire)
Description: The CIS questionnaire was used to assess the parents' sleep. It was completed directly by the parent/carer. The CIS consists of 20 statements on fatigue-related problems responders might have experienced in the past 2 weeks. A Likert scoring scheme from 1 to 7 ranging from 1-"no, that is not true" to 7-"yes, that is true" with items 2, 5, 6, 7, 8, 11, 12, 15 and 20 hold inverted scores. The total score ranges from 20 to 140. The questionnaire covers measures 4 dimensions of fatigue: Subjective fatigue severity (8 items), Concentration problems (5 items), Reduced motivation (4 items) and Physical activity (3 items). Dimensions can be analyzed separately, with higher scores indicating higher levels of subjective fatigue (8-56), reduced concentration (5-35), reduced motivation (4-28), and lower levels of physical activity (3-21). A total score over 76 is considered at risk of a fatigue disorder, while 36 provides the cutoff score on the subjective experience of fatigue sub-scale
Time Frame: Assessment will be done at each study clinic visit (Day 56 +/- 7 )
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DryNites Arm | No Pants Arm
Number analyzed (Participants) | 28 | 61
score on a scale | 43.7 (16.88) | 46.1 (22.75)

ADVERSE EVENTS:
Time Frame: 56 +/- 7 days
Arm/Group | DryNites Arm | No Pants Arm
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/70
Other Adverse Events (participants affected / at risk) | 1/35 | 4/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DryNites Arm (N=35) | No Pants Arm (N=70)
subglottic laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DryNites Arm (N=35) | No Pants Arm (N=70)
genital candidiasis, (Infections and infestations) | 0 (0) | 1 (1)
pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
subglottic laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pyrexia (Infections and infestations) | 0 (0) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04620356/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT04620356/SAP_001.pdf